CLINICAL TRIAL: NCT07307651
Title: Implementation of an RT-PCR Assay for the Diagnosis of Rickettsia Spp. Infection
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Rickettsia2024
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Infection; Rickettsia Infections
MeSH Terms: conditions — Infections; Rickettsia Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective cohort
- prospective cohort

SUMMARY:
Rickettsia2024 is a multicenter, tissue observational, retrospective and prospective cohort study. Enrollment will take place within the outpatient clinics of the Infectious Diseases and Dermatology Unit of the IRCCS AOUBO and, following an infectious disease consultation in the Bologna Metropolitan area, at the Hospitals and CAUs of the Bologna Local Health Authority. Within these UUOOs, biopsy samples from normal clinical practice are performed on patients with strong clinical suspicion of Rickettsia infection: therefore, it will not be necessary to perform any additional samples for the conduct of this study. Samples from the normal diagnostic process are sent to the Microbiology UOC, where they are subjected to various analyses. RT-PCR analyses (commercial or in-house kit) and assay of species-specific IgG antibodies will be performed according to clinical practice. Additional tests will be performed with a commercial kit for retrospective samples and with a home-made method for prospective samples.

DETAILED DESCRIPTION:
It is estimated that a total of approximately 800 patients can be recruited, 400 for the retrospective part and the same number for the prospective part (estimated using data collected from requests received to date). For the retrospective cohort: from January 2023 until approval by the ethics committee; For the prospective cohort: from ethics committee approval until December 2027.

ELIGIBILITY:
Inclusion Criteria:

* pazienti che presentano escara
* pazienti con richiesta del dosaggio degli anticorpi anti-Rickettsia conorii

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients belonging to the UUOOs involved in the study, for whom serum samples, whole blood, skin biopsy, eschar, vesicle buffer underlying the eschar collected through withdrawals that meet the inclusion criteria, performed according to clinical practice, are available:
  * For the retrospective cohort: from January 2023 until approval by the ethics committee;
  * For the prospective cohort: from ethics committee approval until December 2027. The Microbiology Unit is the operational reference unit. The Infectious Diseases and Dermatology Unit of the IRCCS AOUBO is involved in patient enrollment, as are the Hospitals and CAUs of the Bologna Local Health Authority, following requests for infectious disease counseling in the Bologna Metropolitan Area.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2028-06-07 (Estimated); Study Completion 2029-06-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the early diagnostic capability of molecular testing (RT-PCR) for the diagnosis of Rickettsia infection at the time of first blood sampling in suspected cases. | from January 7, 2026 to June 7, 2028

SECONDARY OUTCOMES:
Comparison of the sensitivity and specificity of diagnosis of in-house RT-PCR and commercial kit (Rickettsia spp REAL TIME PCR, Immunospark) | from January 7, 2026 to June 7, 2028
Identification of Rickettsia species by gene sequencing of the 16S rRNA portion of samples tested positive (threshold cycle < 30) by in-house RT-PCR/commercial kit | from January 7, 2026 to June 7, 2028
Estimation of the incidence of Rickettsia conorii infections in the Bologna metropolitan area through serological screening | from January 7, 2026 to June 7, 2028

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - AUSL di Bologna, Bologna, Bologna

REFERENCES:
- [Result] Giulieri S, Jaton K, Cometta A, Trellu LT, Greub G. Development of a duplex real-time PCR for the detection of Rickettsia spp. and typhus group rickettsia in clinical samples. FEMS Immunol Med Microbiol. 2012 Feb;64(1):92-7. doi: 10.1111/j.1574-695X.2011.00910.x. Epub 2011 Dec 12. PMID 22098502
- [Result] Brouqui P, Bacellar F, Baranton G, Birtles RJ, Bjoersdorff A, Blanco JR, Caruso G, Cinco M, Fournier PE, Francavilla E, Jensenius M, Kazar J, Laferl H, Lakos A, Lotric Furlan S, Maurin M, Oteo JA, Parola P, Perez-Eid C, Peter O, Postic D, Raoult D, Tellez A, Tselentis Y, Wilske B; ESCMID Study Group on Coxiella, Anaplasma, Rickettsia and Bartonella; European Network for Surveillance of Tick-Borne Diseases. Guidelines for the diagnosis of tick-borne bacterial diseases in Europe. Clin Microbiol Infect. 2004 Dec;10(12):1108-32. doi: 10.1111/j.1469-0691.2004.01019.x. PMID 15606643
- See also: Related Info — https://www.epicentro.iss.it/zecche/FebbreBottonosa2001-2015
- See also: Related Info — https://doi.org/10.1016/j.ttbdis.2018.09.001